CLINICAL TRIAL: NCT02630927
Title: A Phase I Randomized, Double-blind, Five-Part Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Oral Doses of AG-519, the Relative Bioavailability of Prototype Tablet Formulations Compared With a Suspension Formulation, and to Evaluate the Pharmacokinetics of a Selected Tablet Formulation Under Fed and Fasted Conditions in Healthy Subjects
Brief Title: A Safety and Tolerability Study of AG-519 in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Agios is no longer developing its second pyruvate kinase-R (PKR) activator, AG-519, and withdrew its investigational new drug (IND) application in December 2016
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AG519-C-001
Record Dates: First submitted 2015-12-08; First posted 2015-12-15 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Anemia
Keywords: Safety and Tolerability; Pharmacokinetic Study; Healthy Volunteer; Pyruvate Kinase; Rare Genetic
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1 Single-Ascending (SAD Phase) (Placebo Comparator): A range of doses of AG519 will be tested based on the assessment of safety and tolerability. A single dose of AG-519 will be administered by mouth (orally).
  Interventions: Drug: AG-519; Drug: Placebo
- Part 2 Multiple-Ascending (MAD Phase) (Placebo Comparator): A range of doses of AG519 will be tested based on the assessment of safety and tolerability. AG519 will be administered by mouth (orally) each day for a period up to 14 days.
  Interventions: Drug: AG-519; Drug: Placebo
- Part 3 Bioavailability & Food Effect (Experimental): The dose to be assessed in Part 3 will be selected based on emerging safety, tolerability and PK/PD data from preceding cohorts in Part 1 and Part 2, which will be reviewed during a dose decision meeting.
  Interventions: Drug: AG-519
- Experimental Part 4 (Subjects of Japanese Origin) (Experimental): Two dose levels of AG-519 will be tested based on the assessment of safety and tolerability in preceding cohorts in Part 1, Part 2, and Part 3
  Interventions: Drug: AG-519
- Experimental Part 5 Open-label Multiple-Ascending (MAD) (Experimental): Up to two dose levels of AG-519 will be tested based on the assessment of safety and tolerability in preceding cohorts in Part 1, Part 2, and Part 3. AG519 will be administered by mouth (orally) each day for a period up to 14 days.
  Interventions: Drug: AG-519

INTERVENTIONS:
Drug: AG-519 — AG519 will be tested.
Drug: Placebo — Placebo will be tested.
  Arms: Part 1 Single-Ascending (SAD Phase); Part 2 Multiple-Ascending (MAD Phase)

SUMMARY:
The purpose of the study is to investigate a drug called AG-519, which is being developed for the treatment of a disease called pyruvate kinase deficiency (also known as PK deficiency) and other forms of anemia. This study is a 5 part study with Part 1 enrolling healthy volunteers into single ascending dose (SAD) groups, Part 2 enrolling healthy volunteers into multiple ascending dose (MAD) groups and Part 3 enrolling healthy volunteers to investigate how much of the study drug is taken up by the body and how food affects the uptake of a prototype formulation of AG-519, Part 4 enrolling healthy volunteers of Japanese origin to compare to the results of subjects of non-Japanese origin, and Part 5 a non-randomized, open-label, multiple dose study enrolling healthy volunteers to further investigate how much of the study drug is taken up by the body when dosed over 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female subjects. Female subjects must be of non-childbearing potential.
2. Age 18 to 60 years inclusive at time of consent.
3. Body mass index (BMI) of ≥18.5 to ≤32.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator.
4. Good state of health (mentally and physically) as indicated by a comprehensive clinical assessment (detailed medical history and a complete physical examination), ECG and laboratory investigations.
5. Subjects who are actively non-smokers and have not used other nicotine-containing products for at least 12 months prior to the screening assessment.
6. Must be willing and able to communicate and participate in the whole study.
7. Must provide written informed consent.
8. Must agree to use an adequate method of contraception.
9. Japanese subjects enrolled in Part 4 must be first generation: born in Japan, not having lived outside Japan for 5 to 10 years, able to trace maternal and paternal Japanese ancestry, with no significant change in lifestyle, including diet (at least one Japanese meal consumed per day), since leaving Japan.

Exclusion Criteria:

1. Participation in a clinical research study within the previous 3 months.
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee.
3. Subjects who have previously been enrolled in this study.
4. History of any drug or alcohol abuse in the past 2 years.
5. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine).
6. Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening.
7. Any females of childbearing potential.
8. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening.
9. Subjects who, after 10 min of supine rest, have a systolic blood pressure (BP) ≥140 mmHg (≥150 mmHg in subjects >45 years of age) or a diastolic BP of ≥90 mmHg.
10. Male subjects with QTcF interval (Fridericia's correction factor) ECG >450 msec, or female subjects with QTcF interval ECG >470 msec on screening or Day 1 (pre dose) ECG.
11. Subjects with a history of serious mental illness, that includes, but is not limited to schizophrenia, bipolar disorder, and major depression.
12. Subjects with glucose-6-phosphate-dehydrogenase (G6PD) deficiency.
13. Subjects with a history of any primary malignancy, including a history of melanoma or suspicious undiagnosed skin lesions.
14. Subjects with any other medical or psychological condition, deemed by the investigator to be likely to interfere with a subject's ability to sign informed consent, cooperate, or participate in the study.
15. Subjects who have undergone major surgery within 6 months prior to screening.
16. Clinically significant abnormal biochemistry, hematology or urinalysis as judged by the investigator.
17. Positive drugs of abuse test result at screening or admission.
18. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results.
19. Subjects who are taking, or have taken, any prescribed or over-the-counter drug.
20. Subjects who have used St. John's Wort within 28 days before the first dose of study drug.
21. History of cardiovascular, renal, hepatic, chronic respiratory or GI disease, or hematologic, lymphatic, neurolologic, endocrine, psychiatric, musculoskeletal, genitourinary, immunologic, dermatologic or connective tissue disease or disorders, as judged by the investigator.
22. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients, including history of allergy to sulfonamides.
23. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator.
24. Donation or loss of greater than 400 mL of blood within the previous 3 months.
25. Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 14 days
  Incidence of adverse events and descriptive statistics for safety laboratory parameters, physical exam findings, vital signs and ECGs. This outcome applies to all Parts of the study

SECONDARY OUTCOMES:
Cmax of AG-519 | 4 days (Parts 1, 3, & 4) 17 days (Parts 2 & 5)
  Descriptive statistics will be used to summarize PK parameters of AG-519 for each dose group and, where appropriate, for the entire population. Standard non-compartmental PK parameters will be calculated from individual plasma concentration data.
Tmax of AG-519 | 4 days (Parts 1, 3, & 4) 17 days (Parts 2 & 5)
  Descriptive statistics will be used to summarize PK parameters of AG-519 for each dose group and, where appropriate, for the entire population. Standard non-compartmental PK parameters will be calculated from individual plasma concentration data.
AUC of AG-519 | 4 days (Parts 1, 3, & 4) 17 days (Parts 2 & 5)
  Descriptive statistics will be used to summarize PK parameters of AG-519 for each dose group and, where appropriate, for the entire population. Standard non-compartmental PK parameters will be calculated from individual plasma concentration data.
Change from baseline in whole blood concentration of adenosine triphosphate (ATP) | 4 days (Parts 1 & 3) 17 days (Part 2)
  The potential relationship between AG-519 and metabolic biomarkers will be explored with descriptive and graphical methods.
Change from baseline in whole blood concentration of 2,3 - diphosphoglycerate (2,3-DPG) | 4 days (Parts 1 & 3) 17 days (Part 2)
  The potential relationship between AG-519 and metabolic biomarkers will be explored with descriptive and graphical methods.

CONTACTS AND LOCATIONS:
Overall Officials: Gary A Connor, RN, Study Director — Agios Pharmaceuticals, Inc.
Locations (1):
- Quotient Clinical, Ruddington Fields, Nottingham, United Kingdom